CLINICAL TRIAL: NCT06167733
Title: Safety and Efficacy Assessment of the VERTICA® - a Radio Frequency Device for the Treatment of Erectile Dysfunction
Brief Title: Safety and Efficacy of the VERTICA® RF Device for the Treatment of ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHH-MED Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URN-2022
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Active vs. Sham
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study personnel, including the investigator and raters and study subjects will be blinded to the treatment assignment (active vs. sham)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active (Experimental)
  Interventions: Device: VERTICA Active device
- Sham (Sham Comparator)
  Interventions: Device: VERTICA Sham device

INTERVENTIONS:
Device: VERTICA Active device — VERTICA device with a therapeutic RF energy level
  Arms: Active
Device: VERTICA Sham device — VERTICA device with a low, non-therapeutic RF energy level
  Arms: Sham

SUMMARY:
Adult subjects with mild to moderate and moderate ED who meet the study eligibility criteria will be enrolled in the study. The enrolled subjects will be randomized by a 1:1 ratio to receive the Active or Sham VERTICA® treatment. Baseline assessments will include collection of demographic data, medical history, concomitant medications and baseline clinical examinations. The initial treatment session will be performed in a clinical setting simulating home use to determine proper device use and to evaluate device tolerability, followed by continued home use of the device for a total of 6 months. Patients will be instructed to attempt sexual activity periodically over the course of the study. Every time a sexual intercourse is attempted, the patient will be requested to complete an event log using validated assessments. Patients will present for monthly follow-up visits, during which safety will be evaluated and additional efficacy assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult, heterosexual, males between 22 and 85 years of age
* Subjects diagnosed with organic ED for at least 3 months, according to the American Urology Association (AUA) Guideline Statement 1 (as described in Section 8.1.1 of the study protocol).
* Subjects with an IIEF-EF score between 11-21
* Steady relationship for at least 3 months
* Subject is sexually active, with at least weekly sexual intercourse attempts or 6 times a month
* Subject is willing to sign informed consent and follow study protocol procedures
* Subject has a smartphone

Exclusion Criteria:

* Castrate and late onset hypogonadism
* History of Priapism or Peyronie's Disease
* Surgery or radiotherapy of the pelvic region
* Anatomic penile deformations or penile prosthesis
* Treatment with antiandrogens
* Previous whole gland treatment of the prostate (Cryoablation, HIFU, external beam radiation of seed implantation, Radical prostatectomy any approach, etc.)
* History of urothelial or colorectal cancer
* Major neurological conditions such as Alzheimer's, Parkinson, Multiple sclerosis, ALS, spinal cord injury, pelvic neuropathy
* Evidence of neurogenic bladder or an indwelling Foley catheter or clean intermittent catheterization (CIC) within 30 days
* Subjects who are taking anticoagulation or anti-platelet therapy
* History of psychiatric disorders, premature ejaculation and drug or alcohol abuse
* Subjects who are incarcerated
* Subjects who are cognitively challenged
* Serious heart or lung disease
* Pregnant partner

Ages: 22 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 98 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
A significant difference in the mean change from baseline in the International Index of Erectile Function - Erectile Function domain (IIEF-EF) scores at 12 weeks, between the treatment groups. | 12 weeks
  The IIEF-EF total score ranges between 6 to 30. A higher total score indicates relatively better erectile functioning.
A significant change from baseline in the mean International Index of Erectile Function - Erectile Function domain (IIEF-EF) scores at 12 weeks, within the VERTICA Active treatment group. | 12 weeks
  The IIEF-EF total score ranges between 6 to 30. A higher total score indicates relatively better erectile functioning.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California, Irvine Medical Center, Newport Beach, California
  - San Diego Sexual Medicine, San Diego, California
  - Optimal Health Miami, Aventura, Florida
  - The University of Chicago, Chicago, Illinois
  - Rachel Rubin MD, Bethesda, Maryland
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas